CLINICAL TRIAL: NCT01692652
Title: Changes of Inflammatory Cytokines in the Tears of Moderate and Severe MGD Treated With Topical Loteprednol Etabonate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2012-0463
Record Dates: First submitted 2012-09-17; First posted 2012-09-25 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Moderate and Severe Meibomiang Gland Dysfunction (Stage 3 or Stage 4 Meibomiang Gland Dysfunction)
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lotemax with warm compress group (Experimental): topical loteprednol etabonate (lotemax 0.5%) qid and warm compress & ocular massage (a minimum of four times, once or twice a daily) for 2months
  Interventions: Drug: topical loteprednol etabonate (lotemax 0.5%) with warm compress & ocular massage
- warm compress only group (Active Comparator): warm compress only group
  Interventions: Other: warm compress only group

INTERVENTIONS:
Drug: topical loteprednol etabonate (lotemax 0.5%) with warm compress & ocular massage
  Arms: Lotemax with warm compress group
Other: warm compress only group
  Arms: warm compress only group

SUMMARY:
Meibum lipids are modified in patients with MGD, resulting in tear instability, evaporative dry eye, and eyelid inflammation. These changes add to corneal damages and exacerbate ocular symptoms, which are all associated with the constant release of inflammatory mediators. To our knowledge, there has been no study on tear cytokine levels in MGD patients treated with topical loteprednol etabonate. The investigators, thus, evaluated both inflammatory tear cytokine levels and corresponding clinical outcomes for analyzing the efficacy of topical loteprednol etabonate in moderate and severe MGD. The aim of this research was to determine the concentration of inflammatory tear cytokines in patients with MGD and to compare the changes in tear cytokine levels between topical loteprednol etabonate and warm compress treatment group and warm compress only treatment group.

ELIGIBILITY:
Inclusion Criteria:

(1) stage 3 or 4 meibomian gland dysfunction

Exclusion Criteria:

1. history of previous ocular or intraocular surgery
2. ocular infection, non dry eye ocular inflammation, ocular allergy, autoimmune disease,
3. history of intolerance or hypersensitivity to any component of the study medications,
4. wearing contact lenses during the study period, presence of current punctal occlusion,
5. pregnancy, lactating women, and children.
6. Additionally, patients were excluded if they were using any topical ocular or systemic medication that could be used for the treatment MGD or dry eye, including topical or oral antibiotics, topical cyclosporine A, topical or oral steroids, topical non-steroidal anti-inflammatory drugs, topical ocular allergy medications or artificial tears

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Changes of inflammatory cytokines in the tears of moderate and severe MGD | 1 second before using topical loteprednol etabonate, after 1 month, and after 2 months of using topical loteprednol etabonate
  Cytokines were measured using the BD Cytometric Bead Array (CBA) (BD Bioscience, San Jose, CA). The cytokines analyzedwere IL-6, IL-7, IL-8, IL-1β, IL-17α, MCP-1, TNF-α, IL-12p70, and IFN-γ. Briefly, 20 μL tear fluid was thawed and added to a 50 μL mixture containing each capture antibody-bead reagent and 50 μL detector antibody-phycoerithrin (Ab-PE) reagent. The mixture was subsequently incubated for 3 h at room temperature, and washed to remove unbound detector Ab-PE reagent before flow cytometry. Data were acquired and analyzed using BD CBA software that calculates the cytokine concentration based on the standard curves and a four-parameter logistic curve-fitting model. Flow cytometry was performed using the BDTM LSRII system (BD Bioscience, San Jose, CA).

CONTACTS AND LOCATIONS:
Locations (1):
- department of Ophthalmology, Yonsei University College of Medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Lee H, Chung B, Kim KS, Seo KY, Choi BJ, Kim TI. Effects of topical loteprednol etabonate on tear cytokines and clinical outcomes in moderate and severe meibomian gland dysfunction: randomized clinical trial. Am J Ophthalmol. 2014 Dec;158(6):1172-1183.e1. doi: 10.1016/j.ajo.2014.08.015. Epub 2014 Aug 13. PMID 25128594